CLINICAL TRIAL: NCT04114617
Title: Physiological Flow of Liquids in Healthy Swallowing
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-9431; 5R01DC011020 (NIH); CAPCR 15-9431 (NIH_HV) (Other: UHN Research Ethics Board)
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Deglutition; Healthy Swallowing; Aging
Keywords: Swallowing; Deglutition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: Participants will be asked to swallow a series of up to 54 liquid stimuli: a) liquid barium (different brands and concentrations); b) a 20% w/v concentration liquid barium thickened to different consistencies using either a starch-based or xanthan-gum based food thickener; and c) lemon-flavored water thickened to different consistencies using either a starch-based or xanthan-gum based food thickener.
  Interventions: Other: Starch-thickened liquids; Other: Xanthan-gum thickened liquids; Combination Product: Barium concentration

INTERVENTIONS:
Other: Starch-thickened liquids — Thickener added in amounts required to reach slightly thick, mildly thick, moderately thick and extremely thick consistencies, as defined by the International Dysphagia Diet Standardisation Initiative flow test.
  Other Names: Nestle Resource ThickenUp
Other: Xanthan-gum thickened liquids — Thickener added in amounts required to reach slightly thick, mildly thick, moderately thick and extremely thick consistencies, as defined by the International Dysphagia Diet Standardisation Initiative flow test.
  Other Names: Nestle Resource ThickenUp Clear
Combination Product: Barium concentration — Commercially available barium products diluted to different concentrations (i.e., 20% w/v, 40% w/v) through the addition of water
  Other Names: Bracco E-Z-Paque barium powder; Bracco E-Z-HD barium suspension; Bracco Polibar Plus liquid barium suspension

SUMMARY:
Thickened liquids are commonly used as an intervention for people with dysphagia (swallowing impairment). However, the field currently lacks a proper understanding of how this intervention works. The overall goal of the project is to collect measurements of bolus flow through the oropharynx (i.e., mouth and throat) during swallowing. The factors that are expected to influence bolus flow include the liquid/food consistency (i.e., thin, slightly-thick, mildly-thick, moderately-thick, extremely thick, solid) and the forces applied during swallowing (i.e., tongue pressures and swallowing muscle contraction). The objective is to determine how these factors interact to influence the flow of a bolus through the oropharynx in healthy swallowing.

DETAILED DESCRIPTION:
The aims of this study are as follows:

Aim 1: To determine the relationship between bolus flow and healthy swallowing physiology. The investigators will collect concurrent videofluoroscopic and physiological measures of swallowing (tongue pressure, electromyography [sEMG]) in healthy adults using barium stimuli across the continuum of liquid consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquids, as defined by the International Dysphagia Diet Standardisation Initiative, www.iddsi.org). Significance: This will show the impact of consistency on bolus flow through the oropharynx, controlling for the forces used to initiate flow and propel the bolus.

Aim 2: To compare healthy swallowing physiology for barium versus non-barium stimuli. The investigators will collect physiological measures of swallowing using barium and non-barium stimuli matched for consistency. Significance: This will determine how swallowing behaviors (tongue pressures, sEMG) differ between barium and non-barium stimuli with matched consistency, enabling us to develop models of flow accounting for these differences.

Aim 3: To compare healthy swallowing physiology across different commercial barium products. Significance: This will determine whether differences in barium concentration or brand influence swallowing behaviors, enabling us to make recommendations regarding ideal contrast agents for use in radiographic swallowing assessment.

ELIGIBILITY:
Inclusion Criteria:

- healthy adults

Exclusion Criteria:

* prior history of swallowing, motor speech, gastro-esophageal or neurological difficulties, chronic sinusitis or taste disturbance
* history of surgery to the speech or swallowing apparatus (other than routine tonsillectomy or adenoidectomy)
* Type 1 Diabetes
* cognitive communication difficulties that may hinder comprehension of the study documents
* known allergies to latex, food coloring or dental glue
* current pregnancy
* recent x-ray to the neck (in the past 6 months)
* occupationally exposure to radiation exceeding 10 milliSieverts in the year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Steele, PhD, Principal Investigator — KITE - Toronto Rehabilitation Institute, University Health Network
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Swallowing of Various Consistencies of Liquid Barium: Healthy adults (without any history or complaints of swallowing impairment) were asked to swallow comfortable sips of different consistencies of liquid barium (thin, slightly thick, mildly thick, moderately thick, extremely thick). Consistencies were defined according to the International Dysphagia Diet Standardisation Initiative Framework. Each participant took 3 sips of each consistency and swallowed without a cue from the investigator.
Period: Overall Study
Arm/Group | Healthy Swallowing of Various Consistencies of Liquid Barium
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults with no history of dysphagia or related conditions.
Groups:
- Healthy Adults: Healthy adults aged 18-82.
Arm/Group | Healthy Adults
Number analyzed (Participants) | 80
Age, Continuous [Mean (Full Range); unit: years] | 46 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 61
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unsafe Swallowing
Description: Swallowing safety was measured using the Penetration-Aspiration Scale, an 8-point categorical scale which captures the depth to which any material enters the airway and whether or not the material is ejected. Levels 1 and 2 on the scale are considered safe, while levels > 2 are considered unsafe. Actual scale scores (1-8) will be recorded and then converted to binary categorical scores (< 3 vs >/= 3). We will report the frequency (count) of participants showing scores > 2 by bolus consistency.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due data quality issues, partial data were missing for thin liquid for 4 participants, and for 3 participants for the remaining consistencies.
Measure: Count of Participants; unit: Participants
Groups:
- Thin Liquid Barium: Participants were asked to take a series of 3 comfortably sized sips of thin liquid barium (Bracco E-Z-Paque powder) prepared in a 20% w/v concentration with water, and to swallow each sip when ready (without a cue).
- Slightly Thick Liquid Barium: Participants were asked to take a series of 3 comfortably sized sips of slightly thick barium, prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, bottled water, and Nestle Resource ThickenUp Clear xanthan gum thickener. Participants were instructed to swallow when ready (without a cue).
- Mildly Thick Liquid Barium: Participants were asked to take a series of 3 comfortably sized sips of mildly thick barium, prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, bottled water, and Nestle Resource ThickenUp Clear xanthan gum thickener. Participants were instructed to swallow when ready (without a cue).
- Moderately Thick Liquid Barium: Participants were asked to take a series of 3 comfortably sized boluses of moderately thick barium, prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, bottled water, and Nestle Resource ThickenUp Clear xanthan gum thickener. Participants were instructed to self-administer a comfortable bolus using a teaspoon and swallow when ready (without a cue).
- Extremely Thick Liquid Barium: Participants were asked to take a series of 3 comfortably sized boluses of extremely thick barium, prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, bottled water, and Nestle Resource ThickenUp Clear xanthan gum thickener. Participants were instructed to self-administer a comfortable bolus using a teaspoon and swallow when ready (without a cue).
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
Participants | 7 | 1 | 3 | 0 | 0

2. Primary Outcome: Amount of Residue in the Pharynx
Description: Residue is material remaining behind in the pharynx after the swallow. We measured residue by tracing the area of barium visible on a lateral view x-ray (in pixels, using ImageJ software) and dividing that area by the squared length C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, and enables the comparison of residue severity across different people with different neck length and pharynx size. In healthy swallowing, residue is expected to be minimal. We report median values and 97.5% confidence intervals for amount of residue by consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquids).
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for 4 participants for thin liquid barium and for 3 participants for the remaining consistencies.
Measure: Median (97.5% Confidence Interval); unit: % of the (C2-4)squared scalar reference
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
% of the (C2-4)squared scalar reference | 0.2 [0 to 4.5] | 0.3 [0 to 5.1] | 0.6 [0 to 5.3] | 0.2 [0 to 4.3] | 0.1 [0 to 4.2]

3. Primary Outcome: Number of Participants Displaying More Than 2 Swallows Per Bolus
Description: The number of swallows needed to clear a single bolus will be counted. 1-2 swallows is considered efficient, while > 2 for a single bolus is considered inefficient. We report the frequency (count) of participants displaying > 2 swallows per bolus by consistency.
Time Frame: Baseline (single timepoint only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
Participants | 6 | 2 | 2 | 3 | 3

4. Primary Outcome: Duration of the Time Interval Between the Bolus Entering the Pharynx and Onset of the Pharyngeal Swallow ("Swallow Reaction Time")
Description: The time interval between the first frame showing the bolus entering the pharynx (passing the ramus of the mandible) and the first frame showing onset of the hyoid burst movement in swallowing, calculated in milliseconds. We report median values and 97.5% confidence intervals for each bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid barium). Longer time intervals reflect delays in initiating the pharyngeal swallow.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for 4 participants on thin liquid and for 3 participants on the other consistencies.
Measure: Median (97.5% Confidence Interval); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
milliseconds | 133 [-33 to 967] | 133 [-67 to 934] | 167 [-33 to 1301] | 267 [-67 to 1468] | 367 [-67 to 1701]

5. Primary Outcome: Duration of the Time Interval Between Onset of the Hyoid Burst and Opening of the Upper Esophageal Sphincter
Description: The time interval between the first frame showing onset of the hyoid burst movement in swallowing and the first frame showing opening of the upper esophageal sphincter, calculated in milliseconds. We report median values and 97.5% confidence intervals for each bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid barium). Longer time intervals reflect a delay in opening of the upper esophageal sphincter.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for 4 participants on thin liquid and for 3 participants on the remaining consistencies.
Measure: Median (97.5% Confidence Interval); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
milliseconds | 100 [33 to 200] | 133 [33 to 200] | 133 [33 to 234] | 167 [67 to 267] | 167 [67 to 267]

6. Primary Outcome: Duration of Upper Esophageal Sphincter Opening
Description: The time interval between the first frame showing opening of the upper esophageal sphincter and the first subsequent frame showing closure of the upper esophageal sphincter behind the tail of the bolus, calculated (in milliseconds). We report median values and 97.5% confidence intervals for each bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid barium). Shorter durations of upper esophageal sphincter opening reflect inadequate durations of opening to allow material to pass through the sphincter from the pharynx into the esophagus.
Time Frame: Baseline (single timepoint only)
Population: as for outcome 5
Measure: Median (97.5% Confidence Interval); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
milliseconds | 467 [400 to 634] | 467 [334 to 634] | 467 [334 to 634] | 400 [300 to 534] | 400 [300 to 534]

7. Primary Outcome: Duration of the Time Interval Between Onset of the Pharyngeal Swallow and Closure of the Entrance to the Airway ("Time-to-Laryngeal-Vestibule-Closure")
Description: The time interval between the first frame showing onset of the hyoid burst movement in swallowing and the first frame showing closure of the laryngeal vestibule, calculated in milliseconds. We report median values and 97.5% confidence intervals for each bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid barium). Longer time intervals reflect delays in achieving airway closure.
Time Frame: Baseline (single timepoint only)
Population: as for outcome 5
Measure: Median (97.5% Confidence Interval); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
milliseconds | 133 [33 to 267] | 133 [-100 to 167] | 133 [-33 to 367] | 167 [0 to 300] | 133 [33 to 267]

8. Primary Outcome: Laryngeal Vestibule Closure Duration
Description: The time interval between the first frame showing closure of the entrance to the airway (laryngeal vestibule closure onset) and the first subsequent frame showing opening of the entrance to the airway (laryngeal vestibule closure offset) calculated in milliseconds. We report median values and 97.5% confidence intervals for each bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid barium). Shorter durations of laryngeal vestibule closure reflect premature termination of airway protection.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for 4 participants for thin liquid and for 3 participants for the remaining consistencies.
Measure: Median (97.5% Confidence Interval); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
milliseconds | 467 [300 to 934] | 467 [300 to 767] | 467 [300 to 734] | 434 [300 to 734] | 434 [334 to 634]

9. Primary Outcome: Degree of Pharyngeal Constriction
Description: During swallowing, the muscles of the pharynx contract to achieve constriction (closure) of the pharynx behind the bolus. The squeezing and pressure generated by this action help to move the bolus downwards through the pharynx. We measured the degree of pharyngeal constriction by identifying the frame of greatest pharyngeal constriction, and tracing the area of any unobliterated pharyngeal space on lateral view x-ray (in pixels, using ImageJ software). The resulting area measure was then divided by the squared length of the C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, enabling the comparison of constriction across different people with different neck length and pharynx size. In healthy swallowing, constriction is expected to be complete, with larger measures reflecting incomplete or poor constriction. We report median values and 97.5% confidence intervals for pharyngeal constriction by consistency.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for thin liquid in 4 participants, and for the remaining consistencies in 3 participants.
Measure: Median (97.5% Confidence Interval); unit: % squared C2-C4 cervical spine length
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
% squared C2-C4 cervical spine length | 1 [0 to 6.2] | 1.2 [0 to 5] | 1.2 [0 to 7.5] | 0.7 [0 to 4.9] | 0.2 [0 to 3.8]

10. Primary Outcome: Diameter of Upper Esophageal Sphincter Opening
Description: During swallowing, the upper esophageal sphincter opens to allow the bolus to move from the pharynx into the esophagus. Narrow opening of the sphincter may obstruct bolus flow. We measured the degree (diameter) of upper esophageal sphincter opening on the frame of maximum distension. Line measurements were made in Image J software. This line measure was then divided by the length of the C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, enabling the comparison of constriction across different people with different neck length and pharynx size. We report median values and 97.5% confidence intervals for pharyngeal constriction by consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid).
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data for thin liquid were missing for 4 participants, and for 3 participants on the remaining consistencies.
Measure: Median (97.5% Confidence Interval); unit: % of the C2-C4 Cervical Spine Scalar
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 76 | 77 | 77 | 77 | 77
% of the C2-C4 Cervical Spine Scalar | 21 [9 to 32] | 19 [9 to 31] | 19 [9 to 30] | 15 [8 to 26] | 16 [9 to 26]

11. Primary Outcome: Pharyngeal Area at Rest
Description: The area of the pharynx was measured, in pixels (using ImageJ software), on a lateral view videofluoroscopic image showing the pharynx at rest. The resulting area measure was then divided by the squared length of the C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, enabling the comparison of pharyngeal size across different people with different neck length. Larger pharyngeal area measures may reflect atrophy of the pharyngeal muscles while smaller pharyngeal area may reflect narrowing due to edema.We report median values and 97.5% confidence intervals for pharyngeal area.
Time Frame: Single timepoint (baseline only)
Population: A sample of 80 adults was enrolled. Due to data quality issues, data were missing for 2 participants.
Measure: Median (97.5% Confidence Interval); unit: % of the squared C2-C4 length scalar
Arm/Group | Healthy Adults
Number analyzed (Participants) | 78
% of the squared C2-C4 length scalar | 59 [37 to 92]

12. Secondary Outcome: Amplitude of Tongue-Palate Pressure
Description: During swallowing, the tongue rises to contact the hard palate, generating pressure that squeezes the bolus backwards through the mouth towards the pharynx. The amplitude of tongue-palate pressure were measured continuously throughout swallowing using the KayPentax Digital Swallow Workstation Swallowing Signals Lab 3-bulb tongue pressure array, and the highest (peak) pressure was identified for each swallow. We will report mean values and standard error for peak pressure by bolus consistency (thin, slightly thick, mildly thick and moderately thick liquid). Higher amplitudes of pressure represent greater force for bolus propulsion.
Time Frame: Baseline (single timepoint only)
Population: A sample of 80 adults was enrolled. This parameter was only collected and analyzed in 40 of those participants, aged 21-59. Due to data quality issues, data were missing for 2 participants.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium
Number analyzed (Participants) | 38 | 38 | 38 | 38
mmHg | 16.53 (2.21) | 25.51 (3.58) | 28.61 (3.47) | 51.89 (8.83)

ADVERSE EVENTS:
Time Frame: Within 1 week of data collection
Description: Participants were asked to contact the lab to advise regarding any digestive or other issues experienced after participating in the data collection session. These were reviewed for possible relationship to the study protocol.
Arm/Group | Healthy Adults
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

LIMITATIONS AND CAVEATS:
In a previous submission, we had included 20 adults who participated in a subsequent supplementary experiment exploring chewing, and the number of chews per bolus had been included as a primary outcome measure. These participants did not complete the main experiment described here, therefore they are excluded from this report. A separate protocol has been registered to cover the chewing experiment (NCT05594173).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04114617/Prot_SAP_000.pdf